CLINICAL TRIAL: NCT02135159
Title: A Phase I Study to Evaluate the Feasibility of Different Sequences of Combined Trastuzumab Emtansine (T-DM1) and Whole-brain Radiotherapy in Patients With Brain Metastases From HER2-positive Breast Cancer
Brief Title: Patients With Brain Metastases From HER2-positive Breast Cancer
Acronym: BIRTH
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Institut du Cancer de Montpellier - Val d'Aurelle (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VA2012/38
Record Dates: First submitted 2014-02-06; First posted 2014-05-09 (Estimated); Last update posted 2017-08-14 (Actual); Status verified 2017-08

CONDITIONS: HER2-positive Breast Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- TDM1 concommitant with RT (Experimental): T-DM1 (First injection day 1) followed by brain sequential RT (start day D3), second injection T-DM1 day 22.
  Interventions: Drug: TDM1; Radiation: Brain Sequential RT
- TDM1 during and after RT (Experimental): Brain sequential RT (start day 1) followed by T-DM1 (First injection day 15), second injection T-DM1 day 36.
  Interventions: Drug: TDM1; Radiation: Brain Sequential RT
- RT before TDM1 (Experimental): Brain sequential RT (start day 1) followed by T-DM1 (First injection day 22), second injection T-DM1 day 43.
  Interventions: Drug: TDM1; Radiation: Brain Sequential RT
- TDM1 before RT (Experimental): T-DM1 (First injection day 1) followed by brain sequential and concomitant RT (start day D18), second injection T-DM1 day 22.
  Interventions: Drug: TDM1; Radiation: Brain Sequential RT

INTERVENTIONS:
Drug: TDM1 — administration of the TDM1 by IV perfusion
  Other Names: no other names
Radiation: Brain Sequential RT — local RT
  Other Names: No other names

SUMMARY:
The purpose of this study is to determine the optimal sequences of combined trastuzumab emtansine (T-DM1) and whole-brain radiotherapy in patients presenting brain metastases from HER2-positive breast cancer in terms of acute toxicities and blood/cerebrospinal fluid T-DM1 pharmacokinetics.

DETAILED DESCRIPTION:
Determine the best sequences.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed invasive breast cancer with stage IV disease.
2. HER-2 positive primary tumor, defined as: IHC3+, or IHC2+ and ISH positive.
3. Non operable brain metastases (n ≥ 2) with at least one measurable CNS lesion ≥ 10 mm on T1-weighted gadolinium-enhanced MRI.
4. No stereotaxie radiotherapy indication
5. At least two weeks from any specific breast cancer treatment (such as Trastuzumab, chemotherapy, immunotherapy/biological response modifiers, endocrine therapy and radiotherapy).
6. Adequate hematologic function (ANC ≥1x109/L, platelets ≥100 000/L; Hb >10g/dL), renal function (creatinine ≤ 1.5x UNL) and hepatic function (albumin ≥2.5 g/dL; serum bilirubin ≤1.5x ULN unless due to Gilbert's syndrome; AST and ALT ≤ 5x ULN if documented liver metastasis or ≤ 3x ULN without liver metastasis).
7. At least 18 years old.
8. ECOG Performance Status of 0 to 2.
9. Life expectancy ≥ 3 months.
10. Potentially reproductive patients must agree to use an effective contraceptive method while on treatment, beginning 2 weeks before the first dose of investigational product and for 28 days after the final dose of investigational product for women. Males able to father a child must practice adequate methods of birth control or practice complete abstinence from intercourse from the first dose of investigational treatment until one week after the final dose of investigational treatment.
11. Women of childbearing potential must have a negative serum pregnancy test within 14 days of enrollment and/or urine pregnancy test 48 hours prior to the administration of the first study treatment.
12. Patients must be affiliated to a Social Security System.
13. Patient information and written informed consent form signed.

Exclusion Criteria:

1. Previous whole brain radiotherapy (WBRT) or brain stereotaxie radiotherapy.
2. Planned or concurrent systemic treatment or radiation therapy (other than corticosteroid, bisphosphonates or mannitol).
3. Known contra-indication to MRI.
4. Active concurrent malignancy. If there is a history of prior malignancy, the patient must be disease free for at least 10 years.
5. Patients with other concurrent severe and/or uncontrolled medical disease which could compromise participation in the study, such as :

   * infection,
   * cardiac disease such as uncontrolled hypertension, congestive cardiac failure, ventricular arrhythmias, active ischemic heart disease, myocardial infarction within one year, LVEF ≤ 50%,
   * current active hepatic or renal disease
6. Pregnant women, women who are likely to become pregnant or are breast-feeding.
7. Patients with significantly altered mental status prohibiting the understanding of the study or with psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial.
8. Known hypersensibility to any component of T-DM1
9. Patients who received any other investigational drugs within the 30 days prior to the screening visit.
10. Individual deprived of liberty or placed under the authority of a tutor.
11. Leptomeningeal metastases diagnosed by MRI
12. Inclusion in another protocol within 30 days
13. Brain metastases with severe intracranial hypertension clinical signs
14. Other cancer except the known primary tumor or in situ cervix cancer or basocellular carcinoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2014-02; Primary Completion 2017-02 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
optimal sequences of combined treatment | 3 months
  To determine the optimal sequences of combined trastuzumab emtansine (T-DM1) and whole-brain radiotherapy in patients presenting brain metastases from HER2-positive breast cancer in terms of acute toxicities and blood/cerebrospinal fluid T-DM1 pharmacokinetics.

SECONDARY OUTCOMES:
objective response | 1 year
  Objective responses (complete and partial response) by MRI according to the RECIST criteria (v1.1) and volumetric assessment

CONTACTS AND LOCATIONS:
Overall Officials: David AZRIA, Principal Investigator — ICM Co. Ltd.
Locations (1):
- Institut regional du Cancer - Val d Aurelle, Montpellier, France